CLINICAL TRIAL: NCT03393598
Title: Randomized Multi-centered Study on Enhancement of Autologous Fat Graft Survival by Recipient Site Preparation
Brief Title: Recipient Site Pre-conditioning in Fat Grafting
Acronym: me15Schaefer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Basel, Switzerland (Other)
Collaborators: Clinical Trial Unit, University Hospital Basel, Switzerland (Other); Ospedale Regionale di Lugano (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ch15Schaefer
Record Dates: First submitted 2017-12-12; First posted 2018-01-08 (Actual); Last update posted 2025-03-12 (Actual); Status verified 2025-03

CONDITIONS: Graft Loss; Condition
MeSH Terms: conditions — Disease

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- pre-expansion using Kiwi® VAC-6000M (Experimental): Expansion will be performed using a complete vacuum delivery system called Kiwi® VAC-6000M with the PalmPumpTM (Clinical Innovations, South Murray, Utah, USA).
  Interventions: Device: pre-expansion using Kiwi® VAC-6000M.; Device: pre-expansion-heating
- pre-heating using Hilotherm Calido®. (Experimental): Pre-Heating will be preformed using a Hiloterm Calido® System.
  Interventions: Device: pre-heating using Hilotherm Calido®.; Device: pre-expansion-heating
- pre-expansion-heating (Experimental): Both preconditioning methods Hilotherm Calido® plus Kiwi® VAC-6000M- will be applied.
  Interventions: Device: pre-expansion using Kiwi® VAC-6000M.; Device: pre-heating using Hilotherm Calido®.
- Control (No Intervention): No preconditioning methods will be applied.

INTERVENTIONS:
Device: pre-expansion using Kiwi® VAC-6000M. — The pre-expansion will be performed with Kiwi® VAC-6000M with the PalmPumpTM.
  Arms: pre-expansion using Kiwi® VAC-6000M; pre-expansion-heating
Device: pre-heating using Hilotherm Calido®. — The pre-heating will be performed with Hilotherm Calido®.
  Arms: pre-expansion-heating; pre-heating using Hilotherm Calido®.
Device: pre-expansion-heating — Both preconditioning methods - Kiwi® VAC-6000M and additionally Hilotherm Calido® - will be applied.
  Arms: pre-expansion using Kiwi® VAC-6000M; pre-heating using Hilotherm Calido®.

SUMMARY:
This study aims to investigate the preparation of the recipient site prior to autologous fat grafting (AFG) using different methods.

DETAILED DESCRIPTION:
Autologous fat grafting is emerging as a powerful tool for soft tissue reconstruction and augmentation and is widely used in plastic surgery. However, there is great variability in terms of long-term graft retention (survival). Moreover, the recipient site preparation is the phase of the procedure which received less attention in clinical and pre-clinical investigations. To provide information regarding an effective preparation of the recipient site may potentially lead to improvements in fat graft survival.

ELIGIBILITY:
Inclusion Criteria:

* Informed Consent as documented by signature
* Patients presenting with contracted scars or body contouring deformities, especially as a result of previous radiation therapy or infection, in and around the breast.
* Body mass index superior than 18.5

Exclusion Criteria:

* Need for antiplatelets drugs in the 5 days before surgery and 3 days after,
* Known or suspected non-compliance, drug or alcohol abuse,
* Inability to follow the procedures of the study due to language problems, psychological disorders, dementia of the participant,
* Previous enrolment into the current study,
* Enrolment of the investigator, his or her family members, employees and other dependent persons,
* Patients with haemorrhagic diatheses.

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2018-01-08 (Actual); Primary Completion 2024-04-11 (Actual); Study Completion 2024-04-11 (Actual)

PRIMARY OUTCOMES:
Fat-graft survival volume | 24 (+/-2) weeks after surgery
  percent remaining

SECONDARY OUTCOMES:
POSAS (Patient and Observer Scar Assesment Scale) | day 7 (+/-3), week 12 (+/-2), week 24 (+/-2)
  POSAS includes 2 subscales: Patient Scale and Observer Scale. Both subscales comprise six items scored numerically from 1 to 10. The sum of the two subscales provides the Total Score of the Patient and Observer Scale (minimum score 12, best scar conditions; maximum score 120, worse scar conditions).
Occurence of Site infection | day 7 (+/-3), week 12 (+/-2), week 24 (+/-2)
  An infection of the surgical site according to CDC (Centers for Disease Control and Prevention) has been observed or not observed (yes or no).
Surgical complication rate | day 7 (+/-3), week 12 (+/-2), week 24 (+/-2)
  According to the Dindo-Clavien classification from grade I (any deviation from the normal postoperative course without the need for pharmacological treatment, or surgical endoscopic and radiological intervention) to grade V (death of a patient).
Pain assessed by VAS (Visual Analogue Scale) | day 7 (+/-3), week 12 (+/-2), week 24 (+/-2)
  Patient pain is assessed with VAS (Visual Analogue Scale for Pain) ranging from 0 (no pain) to 10 (worst imaginable pain).

CONTACTS AND LOCATIONS:
Overall Officials: Dirk J Schaefer, Prof MD, Principal Investigator — Plastic, Reconstructive, Aesthetic, and Hand Surgery,
Locations (2):
- Switzerland (2):
  - University Hospital Switzerland, Dept. of plastic, reconstructive, aestetic and hand surgery, Basel
  - Klinik Hirslanden, Plastic Surgery Group AG, Zurich